CLINICAL TRIAL: NCT02077686
Title: A Prospective Multi-center Evaluation of a Diabetes Education Module Specifically Addressing the Topic "Diabetes and Travel" in a Randomized Controlled Trial
Brief Title: Diabetes and Travel: Evaluation of a Diabetes Education Module - a Randomized Controlled Trial (PRIMO_Travel)
Acronym: PRIMO_Travel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, Head of the Research Institut Diabetes Academy Mergentheim, Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH022014_2
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; education; randomized; prospective
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education - Diabetes and Travel (Experimental): Patients randomized to this arm, will participate immediately in the education module "Diabetes and Travel"
  Interventions: Behavioral: Education - Diabetes and Travel
- Waiting-list control group (No Intervention): Patients in the control group will get the education with the education module after completion of the 6-month follow-up

INTERVENTIONS:
Behavioral: Education - Diabetes and Travel — Based on the treatment and education programme PRIMAS a problem-specific education module regarding "Diabetes and Travel" was created. The module covers specific and detailed aspects of the topic "travel" such as insulin adaption to intercontinental flights, dealing with exotic food, and treatment goals during vacation. With this module, a more comprehensive education of patients with specific interest is possible.
  Arms: Education - Diabetes and Travel

SUMMARY:
This study is a multi-center, randomized prospective trial with a 6-month follow up. A newly developed treatment and education module will be tested compared to a waiting-list control group. The module covers the topic "diabetes and travel". Primary outcome variable is diabetes-specific empowerment regarding diabetes and travel. Secondary outcome variables are: diabetes-related distress, health-related quality of life, depressive symptoms, self-care behavior, and glycemic control.

DETAILED DESCRIPTION:
The module consists of one lesson (duration: 90 minutes). The module is derived from the empowerment approach and is based on the previously evaluated education and treatment program for type 1 diabetes: PRIMAS (NCT01220557). The module is designed as a group session held by a trained diabetes educator. Patients are randomized either to the immediate participation in the module or to the control group. Control group is a waiting-list control group. Patients in this waiting-list control group get the education after the completion of the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Intensive insulin treatment
* specific interest in "Diabetes and Travel"
* wish to participate in group education
* informed consent
* fluent in reading and speaking German language

Exclusion Criteria:

* diabetes duration < 4 week
* severe organic disease (e.g. terminal renal disease, cancer with poor prognosis)
* current treatment of a mental disease
* cognitive impairment
* dementia
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2014-02; Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diabetes-specific empowerment on the adapted Diabetes Empowerment Scale at the 2-week and 6-month follow-up | Baseline, 2-week follow-up , 6-month follow-up
  The Diabetes Empowerment Scale was specifically adjusted to cover the topic "travel". Psychometric criteria for these adjusted scale were evaluated in an independent study.

SECONDARY OUTCOMES:
Change from baseline in problem-specific distress on the adapted Problem Areas in Diabetes (PAID) Scale at the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up
  The PAID scale was specifically adapted to cover the topic "travel". Psychometric quality was assessed in an independent study
Change from baseline in glycemic control (HbA1c) at the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up
  HbA1c will be analyzed in a central laboratory.
Change from baseline in health-related quality of life on the EQ-5D at the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up
Change from baseline in quality of life on the WHO-5 at the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up
Change from baseline in self-efficacy on the General Self-Efficacy Scale (GSE) the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up
Change from baseline in general diabetes-distress at the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up
Change from baseline in depressive symptoms on the CES-D at the 2-week and 6-month follow-up | baseline, 2-week follow-up, 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim
Locations (4):
- Germany (4):
  - Research Institute of the Diabetes Academy Mergentheim (FIDAM), Bad Mergentheim
  - Zentrum für Diabetologie Bergedorf, Hamburg
  - Diabeteszentrum Ludwigsburg, Ludwigsburg
  - Diabetologische Schwerpunktpraxis Neuss, Neuss